CLINICAL TRIAL: NCT00341601
Title: A Natural History Study of Multidrug-Resistant Tuberculosis Strains and Host Susceptibility Genes in Korean Patients With Pulmonary Tuberculosis
Brief Title: Multi-Drug Resistant Tuberculosis in Korea
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Tuberculosis Research Center (Other); National Masan Tuberculosis Hospital (Unknown); Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905069; 05-I-N069
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01-29

CONDITIONS: Tuberculosis
Keywords: Mycobacterium Tuberculosis; TLR-2; Recurrent Tuberculosis; Phenolic Glycolipid; mRNA Expression Profiles
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study, conducted in Korea, will examine why some people are more susceptible to tuberculosis (TB) than others and why some strains of M tuberculosis (the bacteria that causes TB) are more difficult to treat or become resistant to drug treatments. The study will compare blood samples and other medical information from patients with different kinds of tuberculosis and with healthy volunteers to identify patient and bacterial characteristics that contribute to disease susceptibility, treatment failure, disease recurrence and multi-drug resistance.

Healthy volunteers and patients with tuberculosis who are 20 years of age or older may be eligible for this study. Subjects are recruited from among patients receiving treatment for tuberculosis at the National Masan Tuberculosis Hospital in the Republic of Korea and from healthy people visiting government health care centers for annual medical checkups. The latter include people who have had TB but are cured; people who have been exposed to TB, but currently have no signs of disease; and those who have not been exposed to TB.

Participants with tuberculosis undergo the following tests and procedures:

* Medical history, including past treatments for TB, and review of medical records
* Interview about home and work
* Sputum collection to test for the kind of TB bacteria present and for genetic studies of the bacteria
* Drug treatment for TB
* Blood draws as part of regular patient care, for HIV testing, and for genetic studies
* Chest x-rays as part of routine patient care
* In patients with recurrent disease, examination of the strains from both bouts of disease to determine if it is a recurrence of the same organism or infection with a new strain.

Healthy volunteers undergo the following tests and procedures:

* Brief medical history
* Blood draw to look for exposure to TB and for genetic studies
* Review of previous x-ray to look for active TB

DETAILED DESCRIPTION:
This natural history study seeks to determine some of the mycobacterial and host factors involved in the failure of antituberculous chemotherapy, disease recurrence, and the development of multidrug resistance by M. tuberculosis. Despite optimal treatment with directly-observed short-course therapy (DOTS), about 5-10% of compliant patients with "cured" tuberculosis relapse, usually within a year after completion of therapy. In Korea, where DOTS is not practiced, the relapse rate has been reported to be 15 to 20 %. In individual patients, failure to eradicate disease contributes directly to the development of drug-resistance and to low overall cure rates. While factors such as patient drug compliance and HIV status have been extensively studied in relation to rates of relapse; host genetic factors and the specific relevance of the infecting mycobacterial strain have not yet been investigated in detail. Identification of patient characteristics and specific strains of M. tuberculosis that are associated with relapse and the evolution of drug resistance would greatly facilitate the development of treatment protocols that might avoid these complications.

Our study population will consist of subjects with pulmonary tuberculosis receiving treatment at our study sites. Healthy volunteers will be selected as the genotypic control population. All subjects with tuberculosis enrolled in the study will be followed by periodic chart review and data extraction during their treatment and follow-up at participating study sites. For 2.5 years after completing drug treatment, tuberculosis recurrence among study subjects will be identified using periodic chart abstraction and follow-up phone calls every 6 months to determine the 2 year recurrence rate for tuberculosis (TB). M. tuberculosis isolates may be collected from subjects with recurrent TB and analyzed to distinguish between relapse and re-infection.

Study subjects will be asked to provide 10 mL of blood and 5 to 30 mL of sputum for acid-fast bacilli (AFB) smear and culture at entry. Sputum will be cultured for M. tuberculosis and isolates will be tested for drug resistance (DR). The research staff may use molecular DR tests to confirm the agar-growth DR results. In addition, subjects will be asked a series of medical history questions including history of prior tuberculosis, antituberculous treatment, disease contacts, and risk factors associated with tuberculosis; and will be asked to give consent to allow clinical research staff to abstract treatment regimens and results from their inpatient and outpatient medical charts for the duration of their participation in the study (treatment and follow-up).

ELIGIBILITY:
* INCLUSION CRITERIA:

For the new cases disease group (Cohort A):

1. Age greater than or equal to 20 years old;
2. Primary treatment (new TB subject by WHO definition) for tuberculosis without treatment interruption (greater than or equal to 60 days) and with at least 4 months of treatment remaining;
3. Clinical signs or symptoms suggestive of tuberculosis;
4. Sputum AFB smear-positivity or confirmed MTB using any molecular test

For previously treated disease group (Cohort B):

1. Age greater than or equal to 20 years old;
2. Treated for tuberculosis previously with more than 30 days of drug treatment and either:

   1. a treatment interruption of greater than or equal to 60 days (includes relapse and treatment after interruption), or
   2. who have experienced treatment failure or have chronic TB.
3. Clinical signs or symptoms suggestive of tuberculosis;
4. Sputum AFB smear-positivity or confirmed MTB using any molecular test

For healthy controls (Cohort C):

1. Age greater than or equal to 20 years old;
2. No previous diagnosis of TB as reported by the subject;

EXCLUSION CRITERIA:

For TB Subjects

1. Women who report themselves to be pregnant or possibly pregnant during the protocol introduction and consent process (pregnant women are not normally treated at NMTH).

For Healthy Volunteers:

1. Women who report themselves to be pregnant or those found to be pregnant by a urine Beta-HCG test during the protocol introduction and consent process.
2. Those having a chest X-ray suggestive of active tuberculosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2005-01-03; Study Completion 2018-01-29

PRIMARY OUTCOMES:
To compare the characteristics of subjects with relapsed tuberculosis verses the characteristics of subjects that do not experience relapse disease | Over course of the study

SECONDARY OUTCOMES:
To compare the frequencies of the Toll-like receptor 2 and 4 (TLR2 and TLR4) alleles in tuberculosis subjects and tuberculosis-exposed, healthy volunteers. Other putative susceptibility genes discussed in the background may also be examined. | End of study
To compare molecular characteristics, including the expression of the phenolic glycolipid, (PGL) of M. tuberculosis strains that occur in subjects with a prior history of disease, disease spread to nonpulmonary sites, or previously treated disea... | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- South Korea (2):
  - National Masan Tuberculosis Hospital & Clinical Research Center, Masan
  - National Medical Center, Seoul

REFERENCES:
- [Background] Abel B, Thieblemont N, Quesniaux VJ, Brown N, Mpagi J, Miyake K, Bihl F, Ryffel B. Toll-like receptor 4 expression is required to control chronic Mycobacterium tuberculosis infection in mice. J Immunol. 2002 Sep 15;169(6):3155-62. doi: 10.4049/jimmunol.169.6.3155. PMID 12218133
- [Background] Acocella G, Conti R. Interaction of rifampicin with other drugs. Tubercle. 1980 Sep;61(3):171-7. doi: 10.1016/0041-3879(80)90007-0. No abstract available. PMID 7003868
- [Background] Agerton T, Valway S, Gore B, Pozsik C, Plikaytis B, Woodley C, Onorato I. Transmission of a highly drug-resistant strain (strain W1) of Mycobacterium tuberculosis. Community outbreak and nosocomial transmission via a contaminated bronchoscope. JAMA. 1997 Oct 1;278(13):1073-7. PMID 9315765
- [Derived] Choi H, Lee M, Chen RY, Kim Y, Yoon S, Joh JS, Park SK, Dodd LE, Lee J, Song T, Cai Y, Goldfeder LC, Via LE, Carroll MW, Barry CE 3rd, Cho SN. Predictors of pulmonary tuberculosis treatment outcomes in South Korea: a prospective cohort study, 2005-2012. BMC Infect Dis. 2014 Jul 2;14:360. doi: 10.1186/1471-2334-14-360. PMID 24990578
- [Derived] Song T, Park Y, Shamputa IC, Seo S, Lee SY, Jeon HS, Choi H, Lee M, Glynne RJ, Barnes SW, Walker JR, Batalov S, Yusim K, Feng S, Tung CS, Theiler J, Via LE, Boshoff HI, Murakami KS, Korber B, Barry CE 3rd, Cho SN. Fitness costs of rifampicin resistance in Mycobacterium tuberculosis are amplified under conditions of nutrient starvation and compensated by mutation in the beta' subunit of RNA polymerase. Mol Microbiol. 2014 Mar;91(6):1106-19. doi: 10.1111/mmi.12520. Epub 2014 Feb 26. PMID 24417450
- [Derived] Cho E, Shamputa IC, Kwak HK, Lee J, Lee M, Hwang S, Jeon D, Kim CT, Cho S, Via LE, Barry CE 3rd, Lee JS. Utility of the REBA MTB-Rifa(R) assay for rapid detection of rifampicin resistant Mycobacterium tuberculosis. BMC Infect Dis. 2013 Oct 15;13:478. doi: 10.1186/1471-2334-13-478. PMID 24128118
- [Derived] Mukundan H, Kumar S, Price DN, Ray SM, Lee YJ, Min S, Eum S, Kubicek-Sutherland J, Resnick JM, Grace WK, Anderson AS, Hwang SH, Cho SN, Via LE, Barry C 3rd, Sakamuri R, Swanson BI. Rapid detection of Mycobacterium tuberculosis biomarkers in a sandwich immunoassay format using a waveguide-based optical biosensor. Tuberculosis (Edinb). 2012 Sep;92(5):407-16. doi: 10.1016/j.tube.2012.05.009. Epub 2012 Jun 17. PMID 22710249